CLINICAL TRIAL: NCT07323511
Title: An Open-Label, Randomized, 8-way Crossover Study to Assess Elements of Abuse Liability of Electronic Nicotine Delivery System Products in Adult Smokers
Brief Title: Abuse Liability for Eight Electronic Nicotine Products
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CSD252101
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Smoking; Smoking Behaviors; Tobacco Use; Tobacco Smoking
MeSH Terms: conditions — Smoking; Tobacco Use; Tobacco Smoking | interventions — HTR3D protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Product usage order ANBGCFDE (Experimental): Subjects will use each of the 8 products during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product N
- Product usage order BACNDGEF (Experimental): Subjects will use each of the 8 products during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product N
- Product usage order CBDAENFG (Experimental): Subjects will use each of the 8 products during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product N
- Product usage order DCEBFAGN (Experimental): Subjects will use each of the 8 products during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product N
- Product usage order EDFCGBNA (Experimental): Subjects will use each of the 8 products during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product N
- Product usage order FEGDNCAB (Experimental): Subjects will use each of the 8 products during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product N
- Product usage order GFNEADBC (Experimental): Subjects will use each of the 8 products during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product N
- Product usage order NGAFBECD (Experimental): Subjects will use each of the 8 products during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product N

INTERVENTIONS:
Other: Product A — Usual Brand (UB) filtered, menthol or non-menthol combustible cigarette
Other: Product B — Tobacco Flavor, 5%
  Other Names: P2815222
Other: Product C — Tobacco Flavor, 1.5%
  Other Names: P2815216
Other: Product D — Tobacco Flavor, 5%
  Other Names: P29156222
Other: Product E — Tobacco Flavor, 2.4%
  Other Names: P2615222
Other: Product F — Tobacco Flavor, 5%
  Other Names: P2615217
Other: Product G — Mint Flavor, 5%
  Other Names: P2915322
Other: Product N — Nicorette® White Ice Mint 4 mg nicotine polacrilex gum

SUMMARY:
This will be a randomized, open-label, 8-way crossover, single-site study designed to evaluate elements of abuse liability (AL), including subjective effects and physiological measures (pharmacodynamics [PD]), and plasma nicotine uptake (pharmacokinetics [PK]) during and following ad libitum use of Electronic Nicotine Delivery System (ENDS) investigational products (IPs) in a confinement setting by generally healthy adult smokers of combustible cigarettes and dual users of cigarettes and ENDS products.

DETAILED DESCRIPTION:
Adult smokers of filtered menthol and/or non-menthol cigarettes and smokers who also use ENDS will be recruited into this study to evaluate elements of ENDS IP AL, in comparison to participant's usual brand (UB) cigarette and nicotine polacrilex gum.

Potential participants will undergo a pre-screening interview followed by a Screening Visit within 28 days prior to enrollment, randomization, and study confinement to assess eligibility.

Eligible participants will be scheduled for a check-in and randomization visit. At this visit, eligibility will be reconfirmed prior to randomization to a product use sequence, based on a Williams design. Participants will then enter a 10-day, 9-night confinement period.

On study Day 1, participants will enter a product familiarization period during which they will be required to use three ENDS IP (Products B,, Product D Product F, and nicotine gum (Product N) at least once. Use of each product during familiarization period will be approximately 5 minutes for each ENDS IP and approximately 30 minutes for a single piece of nicotine gum. After completing this familiarization, they will be permitted to smoke their UB cigarettes ad libitum. Participants who also use other tobacco and/or nicotine-containing products such as ENDS, smokeless tobacco or modern oral nicotine products in addition to their UB cigarettes will not have access to those products during the study.

Following the product familiarization period, participants will enter a product acclimation period (beginning on Day 2 and each day prior to a test session) during which they will use their randomized IP (excluding their UB cigarette) assigned for use in the next day's test session at least four times, for approximately 5 minutes per use for ENDS IPs and approximately 30 minutes for a single piece of nicotine gum use. After completing this requirement, participants will be permitted to smoke their UB cigarettes ad libitum. Pharmacy logs will be used to capture information on product usage during the product familiarization and acclimation periods.

At the end of the product acclimation period and ad libitum use of the participant's UB cigarette, participants will abstain from use of all tobacco- and nicotine-containing products for a minimum of 12 hours prior to each test session occurring on the following day. In addition, participants will be required to abstain from any caffeine-containing products for 4 hours prior to the start of each test session through the end of the test session.

Starting on Day 3 and continuing through Day 10, each participant will participate in eight consecutive daily test sessions, evaluating one IP per session.

Over the course of the study, each participant will evaluate a total of eight IPs:

six ENDS IPs, a high-AL comparator (the participant's UB cigarette), and a low- AL comparator (a commercially available nicotine replacement therapy [NRT] nicotine gum).

During each test session, blood samples will be collected for plasma nicotine PK assessments. Additionally, subjective effects questionnaire responses and physiological measures will be taken before, during, and after each product use.

The active period of each test session will start with assigned IP use initiation and last approximately 4 hours during and following product use. During each test session, participants will be allowed approximately 5 minutes of smoking one UB cigarette; approximately 5 minutes of ENDS IP use; or approximately 30 minutes of nicotine gum use (one piece per package labeling), based on the product use sequence to which participants will be randomized. Participants' use of the ENDS IP will be self-defined during the 5-minute ad libitum IP use session; specific parameters around puff duration, volume, inter puff interval, and quantity will not be prescribed. ENDS IP cartridges will be weighed within 4 hours before and after the test session on Days 3 - 10.

Participant safety will be monitored throughout the study by the Principal Investigator (PI) or qualified designee by adverse events (AEs) assessments, vital sign measurements, physical examinations (including an oral examination), and clinical laboratory tests. The Medical Monitor will be available for consultation throughout the study and for any necessary follow-up after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, understand, and willing to sign an informed consent form (ICF) and complete questionnaires written in English.
* Generally healthy male or female, 21 to 60 years of age, inclusive, at the time of consent.
* Expired breath carbon monoxide level is ≥ 10 ppm and ≤ 100 ppm at Screening.
* Positive (≥200 ng/ml) urine cotinine test at Screening.
* Smokes only combustible filtered, menthol or non-menthol cigarettes, 83 mm to 100 mm in length.
* Agrees to smoke same UB cigarette throughout the study period. UB cigarette is defined as the cigarette brand style currently smoked most frequently by the participant.
* Participants must meet one (a or b) of the following tobacco use conditions:

  1. Smokes at least 10 cigarettes per day (on average) and inhales the smoke, for at least 6 months prior to Screening. Brief periods of abstinence due to illness, quit attempt (more than 30 days prior to Screening), or clinical study participation (more than 30 days prior to Screening) will be allowed at the discretion of the Principal Investigator (PI).
  2. Dual user of cigarettes and ENDS who self-reports:

  i. Smoking at least 10 cigarettes per day (on average) and inhales the smoke, for at least 6 months prior to Screening Visit. Brief periods of abstinence more than 30 days prior to screening due to illness, quit attempt or clinical study participation will be allowed at the discretion of the PI and ii. Using a nicotine-containing ENDS (cartridge or a tank system). NOTE: Cigarette smokers or ENDS users who also use other tobacco- or nicotine-containing products (e.g., smokeless tobacco, and modern oral nicotine products) on no more than one day per week will not be excluded from study participation.
* Response at Screening to the Fagerström Test for Nicotine Dependence (FTND) Question 1 ("How soon after you wake up do you smoke your first cigarette?") is either "Within 5 minutes" or "6-30 minutes."
* Willing to use only UB cigarette, ENDS IPs, and nicotine gum during the study period.
* Willing to abstain from tobacco and nicotine use for at least 12 hours prior to each test session.
* Females must be willing to use a form of contraception acceptable to the PI from the time of signing informed consent until End-of-Study.
* Males must use an acceptable method of birth control from Day 1 "check-in" until the end of the study, unless they have had a vasectomy or are abstinent from heterosexual intercourse, or their female partner is not able to bear children.
* Agrees to in-clinic confinement of 10 days and 9 nights.

Exclusion Criteria:

* Presence of clinically significant uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, gastrointestinal, psychiatric, hematological, neurological disease, or any other concurrent disease or medical condition that, in the opinion of the PI, makes the study participant unsuitable to participate in this clinical study.
* History, presence of, or clinical laboratory test results indicating diabetes.
* Systolic blood pressure of > 160 mmHg or a diastolic blood pressure of > 95 mmHg, measured after being seated for five minutes at Screening and at check-in Day 1.
* Weight of ≤ 110 pounds at Screening.
* Hemoglobin level is < 12.5 g/dL for females or <13.0 g/dL for males at Screening.
* Scheduled treatment for asthma currently or within the past consecutive 12 months prior to the Screening Visit. As-needed treatment, such as inhalers, may be included at the PI's discretion.
* Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
* Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that has been surgically and/or cryogenically removed.
* Must not be a current regular user (i.e., > 5 times per month) of any tobacco products other than cigarettes or ENDS within the last 6 months prior to screening.
* Use of any medication or substance that aids in smoking cessation, including but not limited to any NRT (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), GLP-1 agonists (e.g., Wegovy®, Mounjaro®, and Ozempic®), or lobelia extract within ≤ 30 days prior to the signing of informed consent.
* History or presence of bleeding or clotting disorders.
* Use of daily aspirin (≥ 325 mg) or other daily anticoagulants.
* Whole blood donation within 8 weeks (≤ 56 days) prior to the signing of informed consent and between Screening and check-in Day 1.

NOTE: Participants will be advised against scheduling a whole blood donation for at least 7 days following study completion.

• Plasma donation within ≤ 7 days prior to the signing of informed consent and between Screening and check-in Day 1.

NOTE: Participants will be advised against scheduling a plasma donation for at least 7 days following study completion.

* Participation in another clinical trial within ≤ 30 days prior to the signing of informed consent. The 30-day window for each participant will be derived from the date of the last study event in the previous study to the time of signing the ICF in the current study.
* Females who have a positive pregnancy test at Screening or check-in on Day 1, are pregnant, breastfeeding, or intend to become pregnant during the course of the study.
* Individuals ≥ 35 years of age currently using systemic, estrogen-containing contraception or hormone replacement therapy.
* A positive drug screen without evidence of prescribed corresponding concomitant medication(s) at Screening or Day 1.
* Postpones a decision to quit using tobacco- or nicotine-containing products in order to participate in this study or a previous quit attempt within ≤ 30 days prior to the signing of the ICF.
* Has a significant history of alcoholism or drug abuse within 24 months prior to Screening, as determined by the PI, or has a positive alcohol test at Screening or check-in on Day 1.
* Employed by a tobacco or nicotine company, the study site, or handles tobacco- or nicotine-containing products as part of their job.
* Individuals or their family members that have ongoing litigation with tobacco company(ies).
* Determined by the PI to be inappropriate for this study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
AUECPL 3-240 | 3 minutes to 240 minutes
  area under the effect curve (AUEC) for PL (VAS score-versus-time)
Emax PL | 240 minutes
  maximum effect (maximum PL VAS score after the start of IP use)

CONTACTS AND LOCATIONS:
Overall Officials: Milly Kanobe, Study Director — Reynolds American

IPD SHARING:
Plan to Share IPD: No